CLINICAL TRIAL: NCT02572180
Title: A Biofeedback Training in Schoolchildren With an Attention-Deficit/Hyperactivity Disorder (ADHD): Differential Effects of Training in a 2D or 3D Environment
Brief Title: A Biofeedback Training in Schoolchildren With an Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Ann-Christine Ehlis, Wissenschaftliche Leiterin der Arbeitsgruppe Psychophysiologie und Optische Bildgebung, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEAD_BluHud_524
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Attention-deficit Hyperactivity Disorder of Childhood or Adolescence Nos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NIRS-based NF in 3D (Active Comparator): A near-infrared spectroscopy (NIRS)-based neurofeedback training in which participants learn to increase the BOLD signal in prefrontal cortical regions will take place in a 3D virtual reality classroom environment.
  Interventions: Behavioral: NIRS-based neurofeedback training
- NIRS-based NF in 2D (Active Comparator): A near-infrared spectroscopy (NIRS)-based neurofeedback training in which participants learn to increase the BOLD signal in prefrontal cortical regions will take place in a 2D (normal computer screen) classroom environment.
  Interventions: Behavioral: NIRS-based neurofeedback training
- EMG-based BF in 3D (Active Comparator): An electromyogram (EMG)-based biofeedback training in which participants learn to self-regulate activity of the musculi supraspinatus will take place in a 3D virtual reality classroom environment.
  Interventions: Behavioral: EMG-based biofeedback training

INTERVENTIONS:
Behavioral: EMG-based biofeedback training
  Arms: EMG-based BF in 3D
Behavioral: NIRS-based neurofeedback training
  Arms: NIRS-based NF in 2D; NIRS-based NF in 3D

SUMMARY:
This study aims towards investigating the efficacy of a near-infrared spectroscopy (NIRS)-based neurofeedback training in a virtual reality (VR) classroom in schoolchildren with attention-deficit/hyperactivity disorder (ADHD). The investigators are especially interested in the training's impact on academic performance, executive functioning (EF) and behavioral ADHD symptoms. Furthermore, the investigators aim at examining the influence of teachers' instructional behavior on children with ADHD's learning in a short virtual reality classroom scenario. Several studies provide evidence that poor academic achievement in ADHD is mainly due to impairments in EF and ADHD behavior (e.g., Frazier, Youngstrom, Glutting, & Watkins, 2007; Miller et al., 2013). Furthermore, studies show that these factors are related to neurophysiological characteristics found in electroencephalographic (EEG) or functional NIRS (fNIRS) examinations (e.g., Barry, Clarke, & Johnstone, 2003; Barry, Johnstone, & Clarke, 2003; Loo & Barkley, 2005; Negoro et al., 2010). Neurofeedback trainings aim at improving these neurophysiological as well as cognitive-behavioral deficits (Gevensleben, Moll, Rothenberger, & Heinrich, 2014), and are expected to improve academic performance in children with ADHD accordingly. Training in a VR classroom, from the investigators' perspective, facilitates generalization of self-regulation competences to real-life academic situations and at the same time increases the effort invested into the training compared to a training in 2D settings. Consequently, training in a VR classroom is hypothesized to lead to greater improvement in academic performance, EF and a greater decrease of ADHD symptoms than a training in a 2D setting. Moreover, the investigators hypothesize that these effects are more pronounced in children who receive a NIRS-based neurofeedback training compared to children receiving a biofeedback training based on an electromyogram (EMG).

DETAILED DESCRIPTION:
1. Strategies 90 schoolchildren from Grade 1 to 4 that meet criteria for a DSM-V diagnosis of ADHD (any presentation) will be recruited. The design will involve three groups (n = 30 per group; N = 90) to which recruited children will be assigned randomly, but matched for age, gender, and medication. In addition to VR NIRS NF and VR EMG biofeedback groups, a third group will experience the NIRS NF in the exact same 2D classroom environment.
2. The Study 2.1. Testing Protocol Informed consent discussion: Parents of children pre-diagnosed with ADHD will not undergo a screening process. However, parents whose children have not been pre-diagnosed with ADHD before, will be provided with the German version of the Conners-3 parent ADHD-Index (C3-AI). Only if the screening indicates that the child is at an increased risk of having ADHD, will the investigators proceed with an informed consent discussion. If the screening indicates that it is unlikely that the child has ADHD, the investigators will exclude the child from the study. After the meeting, if the child was either pre-diagnosed with ADHD before, or the screening indicates an increased likelihood for the child to have ADHD, parents will have enough time to think about whether they want to give written informed consent to participate in the study.

If parents give written informed consent, the next step will be a session in which the ADHD diagnosis is verified. For this session, parents will be informed about three opportunities.

1. Diagnostic session in the scope of their participation in a second study at the pediatric clinic in Tübingen at the same time that they participate in our biofeedback study. This study is called "Aufmerksamkeit und Kognition bei Kindern mit Neurofibromatose Typ 1", which is still searching for children with ADHD only (without neurofibromatosis type 1) to form a control group.
2. Diagnostic session in the scope of the "Spezialsprechstunde ADHS" in the outpatient clinic of the department of child and adolescence psychiatry.
3. Diagnostic session within the scope of this biofeedback study as described below.

Diagnostic session: For a standardized confirmation as well as a characterization of the diagnosis, the long versions of the Conners-3 parent and teacher rating scales (3-P and 3-T) will be applied. Furthermore, the German version of the Strengths- and Difficulties Questionnaire (SDQ-Deu) is going to assess the severity of the symptoms as well as comorbidities from class teacher as well as parental perspective. In order to assess the actual quality of life of parents and child parents and children will be asked to fill out the Kiddy-Kindl in its appropriate version. Moreover, surrounding variables such as medication, prior treatment, other clinical diagnoses etc. will be assessed with a questionnaire. As neuropsychological variables, intelligence will be assessed using the short version of the Culture Fair Test (CFT 1-R or CFT 20-R).

Pre-Test:

Session 1 of the pre-test is going to assess executive functions of the participants and requires a washout of methylphenidate (MPH) as well as amphetamines. MPH and amphetamines should be washed out for at least 48 hours over the weekend so that the pre-test can take place on Mondays. Atomoxetine does not need any washout as the effects of medication are not directly related to the drug level in the blood. In this first session, a combined EEG/NIRS-measurement will take place as the investigators would like to provide information about whether changes caused by the BF intervention are also reflected in changes that can be measured with EEG and NIRS during the following tasks: a Go/No-Go Task (10 min.), a verbal fluency task (10 min.) and an n-back task (10 min.). Furthermore, the participants' performance on a digit span task (forward & backward) (10 min.) will assess verbal WM whereas a matrices span task (15 min.) and the Corsi Block Tapping Task (forward & backward) (10 min.) will assess visual-spatial WM performance. Inhibition will be once more assessed using the Stop Signal Task (10 min.).

Session 2 (without medication washout) will assess academic performance using one of the appropriate DEMAT 1+-4 (20-40 Min.) assessing mathematical performance and the SLRT-II (25-35 Min.) assessing reading and writing performance. Furthermore, sustained attention will be assessed with the Conner's CPT (15 min.). Questionnaires assessing self-control and academic self-efficacy will be filled out by the children (ca. 20 min.).

Furthermore, an accelerometer that is worn on the non-dominant side of the body (hip), attached to the waistband with a light belt, for ten consecutive days will objectively assess motor hyperactivity. During this time, parents will be called once per day to assess ADHD symptoms with the Global Index ADHD (ADHS-GI) and to check whether the accelerometer is worn and works.

Parents and teachers will be asked to fill out the BRIEF as well as the SDQ-Deu, the long versions of the Conners-3 parent and teacher rating scales (3-P and 3-T) and the Kiddy-Kindl. Moreover, the investigators will ask the parents to fill out an adapted version of the FERT as well as an adapted version of the brief self-control scale in order to assess their expectancies of the training.

Midway-Test: After eight sessions, participants will have a break of two to three weeks in which no NF or BF training takes place. ADHD behavior will be assessed by asking parents as well as teachers to fill out the Conners 3-P/ 3-T.

Post-Test: The post-test will follow the procedure already applied in the pre-test.

Follow-Up-Test (6 months after the last training session): The Follow-Up-Test will follow the course of the post-test exactly.

Every session. During every session, the investigators will assess the participant's motivation with a short questionnaire measuring joy, effort and enthusiasm. Furthermore, heart rate variability (HRV) will be recorded as it has been shown to be related to motivational processes. Accelerometer data from knee and wrist will be recorded to examine hyperactive behavior.

2.2. Training Plan and Protocol The NIRS- and EMG-based NF and BF training protocols of this study will include 15 training sessions in total, two to three per week. Every training session will last about 60 minutes including the biofeedback training itself and a preparation phase at the beginning, in which the NIRS cap and its optodes are fitted to the head in the case of a NF training, or the EMG electrodes are placed above both Musculi supraspinatus in the case of a BF training. Furthermore, the head-mounted display (HMD) for the VR is mounted (in the VR 3D classroom groups only).

Every training session with NIRS- and EMG-based NF/BF consists of three runs, of which the first and the second are with continuous performance feedback (feedback condition). In the third run, no feedback is provided (transfer condition). Lighting in the 3D VR or 2D classroom increases with activation and decreases with deactivation. During the first eight training sessions, the training will follow a protocol with 50% activation and 50% deactivation trials. For the second half of the training sessions, the protocol will change to 80% activation and 20% deactivation trials.

After eight sessions, participants will have a two to three week break that aims at further supporting transfer to a real-life setting by using stimulus cards with screenshots of the training setting and instructions to practice activation and deactivation at home on a daily basis. The stimulus cards show the image of the classroom participants see during the training and will be introduced in the laboratory setting directly after the training sessions 6, 7 and 8. That means, with the help of these cards and while looking at them, participants should practice brain or muscular activation several times (depending on whether they belong to the NIRS-NF or EMG-BF group) like they learned in the training, i.e. they should imagine to increase the lighting in the room when looking at the stimulus cards for two to four minutes. After this activation task, they solve some mathematical tasks or riddles matching their age and knowledge. In the second half of the training sessions, after the break, participants are asked to continue practicing activation at home before doing their homework as well as in other situations requiring attention.

2.3. Experimental Paradigm Participants that receive a NIRS-based NF training have to increase the BOLD signal (activation) or decrease it accordingly (deactivation). Analogously, participants in the BF training condition will have to increase and decrease muscular activity measured with EMG. Every session consists of three runs. In the first and the second run, contingent performance feedback is provided, but no feedback is given in the third run. Feedback will be provided to the participants via a continuous change of the lighting within the room; the room will brighten with increasing activation and dim with increasing deactivation. Additional feedback from an animated teacher as well as a scoreboard will provide them with positive reinforcement at the end of every trial.

Visual, auditory and mixed distractors such as, for instance, paper planes flying through the room, fellow students whispering, or people knocking on the door and coming into the room, will be introduced in every run from the fourth training session onwards. The distractors appear with a distance of at least 60 seconds between two distractors.

The baseline of the first, second and third run will be calculated from the BOLD signal in the last two seconds before the trigger (arrow) appears. Reinforcement will be provided with 1 smiley when the participant spent 60% of the time of the second half of the trial on the required side of the baseline (i.e., below, if deactivation is required, or above, if activation is required). Analogously he/ she will receive 2 smileys with 70% and 3 smileys with 80% of the second half of the trial in the required direction. Reinforcement for the second run changes adaptively with the performance in the first run. If the participant scored between 40-60 % success rate (getting at least 1 smiley), the second block will remain exactly like the first. If the participant scores lower than 40% success rate, the threshold will decrease to 0.8 standard deviations (STD) in either direction relative to the baseline, so that the normalization of the light makes it more sensitive to performance. In addition, the threshold for getting a smiley would decrease to 50%, 60%, and 70% for one, two or three smileys respectively. If the participant scores higher than 60 % success rate in the first run, then the threshold would increase to 1.2 STD above and below the baseline. In addition, the percent of time that is spent above the baseline or below the baseline would need to be 0.1 STD above or below the baseline to count towards the overall percentage. The third run is the same as the second in calculation.

ELIGIBILITY:
Inclusion Criteria:

* Going to school Grade 1-4.
* Clinical diagnosis of ADHD combined, predominantly inattentive or predominantly hyperactive-impulsive type according to DSM-V.
* IQ > 70 as assessed with the CFT 1-R or CFT 20-R (Weiß & Osterland, 2013; Weiß & Weiß, 2006).
* No additional serious physical, neurological or mental disorder as specified below.

Exclusion Criteria:

* Not going to school or in other Grades than 1-4.
* No clinical diagnosis of ADHD according to the DSM-V.
* IQ < 70 as assessed with the CFT 1-R or CFT 20-R (Weiß & Osterland, 2013; Weiß & Weiß, 2006).
* Parent reported diagnosis of the following: Serious physical illness or chronic diseases such as lung disease, heart disease, diabetes, hypertension, and rheumatic diseases; Neurological disorders including stroke, multiple sclerosis and epilepsy; indicated psychiatric disorders including obsessive-compulsive disorder, chronic tics, Tourette syndrome, and suicidal behavior.
* Prior participation in a BF/NF training.
* Other psychotherapeutic treatment or any kind of attention training, also in the course of an ergotherapeutic treatment, while participating in the study.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
ADHD symptomatology | 9 months
  ADHD symptomatology will be measured as evaluated by teachers and parents using the German long version of the Conners-3. Furthermore, data from accelerometer measures will provide information about motor hyperactivity. The SDQ and the KINDL will assess the children's and family's quality of life which is directly associated with ADHD symptomatology.
Activity in diverse cortical regions and parallel behavioral performance | 9 months
  The investigators measure prefrontal cortical activity using near-infrared spectroscopy and electroencephalography (EEG) during the verbal fluency task, the Go/NoGo and the n-back task. Behavioral performance on these tasks will also be assessed.

SECONDARY OUTCOMES:
Executive functions | 9 months
  Using a variety of neuropsychological tests, the investigators aim at testing executive functioning using a digit span task, a matrices span task, the corsi block tapping task, and the stop signal task. Furthermore, parents and teachers will evaluate executive functioning with the BRIEF.
Academic performance | 9 months
  Academic performance in math and German will be assessed using an age-appropriate version of the LVD-M 2-4 and the SLRT-II.
Sustained attention | 9 months
  Sustained attention will be measured using the Conner's continuous performance task (CPT).
Self-control and academic self-efficacy | 9 months
  These variables are assessed using adapted versions of the following questionnaires:
  1. Brief version of the self-control scale (for parents and children)
  2. Questionnaire on academic self-efficacy
Expectations of parents | 9 months
  The expectations of parents on the bio- and neurofeedback interventions will be assessed using an adapted version of the FERT.
Motivation for the intervention | 3-4 months
  Motivation of the participants for the intervention will be assessed directly before every training session starts using a short self-assessment mainkin. Furthermore, an electrocardiogram (ECG) allows the investigators to measure the heart-rate variability which is hypothesized to be directly associated with motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Christine Ehlis, Dr., Principal Investigator — Psychiatry and Psychotherapy (Uni Tübingen); Caterina Gawrilow, Prof., Principal Investigator — School Psychology (Uni Tübingen); Thomas Dresler, Dr., Principal Investigator — LEAD Graduate School; Tobias J Renner, Prof., Principal Investigator — Child and Adolescence Psychiatry (Uni Tübingen)
Locations (1):
- LEAD Graduate School, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. (2013). DSM-5 Attention Deficit/ Hyperactivity Disorder Fact Sheet. American Psychiatric Association. Retrieved from www.dsm5.org
- [Background] Arns M, de Ridder S, Strehl U, Breteler M, Coenen A. Efficacy of neurofeedback treatment in ADHD: the effects on inattention, impulsivity and hyperactivity: a meta-analysis. Clin EEG Neurosci. 2009 Jul;40(3):180-9. doi: 10.1177/155005940904000311. PMID 19715181
- [Background] Barry RJ, Clarke AR, Johnstone SJ. A review of electrophysiology in attention-deficit/hyperactivity disorder: I. Qualitative and quantitative electroencephalography. Clin Neurophysiol. 2003 Feb;114(2):171-83. doi: 10.1016/s1388-2457(02)00362-0. PMID 12559224
- [Background] Barry RJ, Johnstone SJ, Clarke AR. A review of electrophysiology in attention-deficit/hyperactivity disorder: II. Event-related potentials. Clin Neurophysiol. 2003 Feb;114(2):184-98. doi: 10.1016/s1388-2457(02)00363-2. PMID 12559225
- [Background] Bertrams, A., & Dickhäuser, O. (2009). Messung dispositioneller Selbstkontroll-Kapazität. Diagnostica, 55(1), 2-10. doi:10.1026/0012-1924.55.1.2
- [Background] Borger N, van der Meere J, Ronner A, Alberts E, Geuze R, Bogte H. Heart rate variability and sustained attention in ADHD children. J Abnorm Child Psychol. 1999 Feb;27(1):25-33. doi: 10.1023/a:1022610306984. PMID 10197404
- [Background] Corsi, P. M. (1973). Human Memory and the Medial Temporal Region of the Brain. Dissertation Abstracts International, 34(2-B), 891.
- [Background] Drechsler, R., & Steinhausen, H.-C. (2013). BRIEF. Verhaltensinventar zur Beurteilung exekutiver Funktionen. Göttingen: Hogrefe Verlag.
- [Background] Drechsler R, Straub M, Doehnert M, Heinrich H, Steinhausen HC, Brandeis D. 1Controlled evaluation of a neurofeedback training of slow cortical potentials in children with Attention Deficit/Hyperactivity Disorder (ADHD). Behav Brain Funct. 2007 Jul 26;3:35. doi: 10.1186/1744-9081-3-35. PMID 17655749
- [Background] Ehlis AC, Bahne CG, Jacob CP, Herrmann MJ, Fallgatter AJ. Reduced lateral prefrontal activation in adult patients with attention-deficit/hyperactivity disorder (ADHD) during a working memory task: a functional near-infrared spectroscopy (fNIRS) study. J Psychiatr Res. 2008 Oct;42(13):1060-7. doi: 10.1016/j.jpsychires.2007.11.011. Epub 2008 Jan 28. PMID 18226818
- [Background] Gevensleben H, Moll GH, Rothenberger A, Heinrich H. Neurofeedback in attention-deficit/hyperactivity disorder - different models, different ways of application. Front Hum Neurosci. 2014 Oct 21;8:846. doi: 10.3389/fnhum.2014.00846. eCollection 2014. PMID 25374528
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Lidzba, K., Christiansen, H., & Drechsler, R. (2013). Conners Skalen zu Aufmerksamkeit und Verhalten-3. Deutschsprachige Adaption der Conners 3rd edition von Keith Conners. Bern: Huber.
- [Background] Marx AM, Ehlis AC, Furdea A, Holtmann M, Banaschewski T, Brandeis D, Rothenberger A, Gevensleben H, Freitag CM, Fuchsenberger Y, Fallgatter AJ, Strehl U. Near-infrared spectroscopy (NIRS) neurofeedback as a treatment for children with attention deficit hyperactivity disorder (ADHD)-a pilot study. Front Hum Neurosci. 2015 Jan 7;8:1038. doi: 10.3389/fnhum.2014.01038. eCollection 2014. PMID 25610390
- [Background] Moll, K., & Landerl, K. (2014). Lese- und Rechtschreibtest (SLRT-II). Weiterentwicklung des Salzburger Lese- und Rechtschreibtests (SLRT) (2., korrig.). Bern: Verlag Hans Huber.
- [Background] Negoro H, Sawada M, Iida J, Ota T, Tanaka S, Kishimoto T. Prefrontal dysfunction in attention-deficit/hyperactivity disorder as measured by near-infrared spectroscopy. Child Psychiatry Hum Dev. 2010 Apr;41(2):193-203. doi: 10.1007/s10578-009-0160-y. PMID 19826946
- [Background] Ravens-Sieberer U, Bullinger M. Assessing health-related quality of life in chronically ill children with the German KINDL: first psychometric and content analytical results. Qual Life Res. 1998 Jul;7(5):399-407. doi: 10.1023/a:1008853819715. PMID 9691720
- [Background] Schwarzer, R., & Jerusalem, M. (1999). Skalen zur Erfassung von Lehrer-und Schüler-merkmalen. Dokumentation der psychometrischen Verfahren im Rahmen der Wissenschaftlichen Begleitung des Modellversuchs Selbstwirksame Schulen. Berlin.
- [Background] Verbruggen F, Logan GD, Stevens MA. STOP-IT: Windows executable software for the stop-signal paradigm. Behav Res Methods. 2008 May;40(2):479-83. doi: 10.3758/brm.40.2.479. PMID 18522058
- [Background] Verbruggen, F., Logan, G. D., & Stevens, M. A. (2013). STOP-IT. Retrieved from http://www.psy.vanderbilt.edu/faculty/logan/#stopit
- [Background] Vollmann, K., Hautzinger, M., & Strehl, U. (2009). Entwicklung und Überprüfung eines Fragebogens zur Erfassung relevanter Therapiebedingungen (FERT) [dissertation]. Tübingen (Deutschland): Eberhard-Karls-Universität Tübingen.
- [Background] Weiß, R. H., & Osterland, J. (2013). CFT 1-R. Grundintelligenztest Skala 1 - Revision -. Göttingen: Hogrefe Verlag.
- [Background] Weiß, R. H., & Weiß, B. (2006). CFT 20-R. Grundintelligenztest Skala 2 - Revision -. Göttingen: Hogrefe Verlag.
- [Background] Conners, C. K., & Sitarenios, G. (2011). Conners' Continuous Performance Test (CPT). In J. Kreutzer, J. DeLuca, & B. Caplan (Eds.), Encyclopedia of Clinical Neuropsychology SE - 1535 (pp. 681-683). Springer New York. doi:10.1007/978-0-387-79948-3_1535
- [Background] Strathmann, A. M., & Klauer, K. J. (2012). LVD-M 2-4 Lernverlaufsdiagnostik für zweite bis vierte Klassen. Göttingen: Hogrefe.
- [Derived] Blume F, Hudak J, Dresler T, Ehlis AC, Kuhnhausen J, Renner TJ, Gawrilow C. NIRS-based neurofeedback training in a virtual reality classroom for children with attention-deficit/hyperactivity disorder: study protocol for a randomized controlled trial. Trials. 2017 Jan 24;18(1):41. doi: 10.1186/s13063-016-1769-3. PMID 28118856